CLINICAL TRIAL: NCT04645875
Title: Effects of Substituting Sitting With Standing and Light Intensity Activity in Free-living Conditions on Glycaemia in Overweight and Obese South Asian Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bedfordshire (Other)
Responsible Party: Principal Investigator, KAMALESH DEY, PhD Candidate, University of Bedfordshire
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2020ISPAR006
Record Dates: First submitted 2020-11-19; First posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Cardiovascular Risk Factor; Cardiovascular Diseases; Diabetes; Type 2 Diabetes; Sedentary Behavior; Sedentary Lifestyle
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Diabetes Mellitus, Type 2; Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sit regimen (Experimental): Participants will be instructed to restrict walking and standing to ≤1 h/day each (total ≤2 h/day ) and the remainder of the waking day will be seated apart from visiting the toilet.
  Interventions: Other: Sit regimen
- SitLess regimen (Experimental): Participants will be instructed to substitute a minimum of 5h/day of sitting with ≥2 h of light-intensity physical activity and ≥3 h of standing. Participants will be advised to rise from the seated position for 2-5 min every 30 min to engage in standing /light-intensity physical activities to interrupt their sitting.
  Interventions: Other: SitLess regimen

INTERVENTIONS:
Other: Sit regimen — See Sit regimen arm description
  Arms: Sit regimen
Other: SitLess regimen — See SitLess regimen arm description
  Arms: SitLess regimen

SUMMARY:
The purpose of this study is to examine whether substituting sitting with standing and light-intensity activity in free-living conditions can reduce glycaemia in overweight/obese South Asian adults.

DETAILED DESCRIPTION:
Anthropometric measurement tools including a stadiometer, a measurement tape and digital weighing scale, activity monitor and Flash Glucose Monitor and sensor will be posted to the participants' home or workplace or research team drop all these items to participants' doorstep to allow participants to take their measures including height, weight, and waist circumference.

Every participant will have to perform a try-out day of the SitLess regimen for 24 hours before starting the study and it will be performed after preliminary testing and before the first experimental condition. Those participants will be included for this study who will be able to adhere to the protocol based on a review of the activPAL activity monitor data that will be worn during the day. Additionally, a second attempt will be offered to them to adhere to the protocol if needed.

Participants will undertake two separate activity regimens in free-living conditions which will be lasting 4-day each condition in a random order:

# Sit regimen: Participants will be instructed to restrict walking and standing to ≤1 h/day each (total ≤2 h/day ) and the remainder of the waking day will be seated apart from visiting the toilet. They will be allowed to perform their daily activities including cooking and other household activities within the 2 h of permitted walking and standing.

#SitLess regimen: Participants will be instructed to substitute a minimum of 5h/day of sitting with ≥2 h of light-intensity physical activity and ≥3 h of standing. Participants will be advised to rise from the seated position for 2-5 min every 30 min to engage in standing /light-intensity physical activities to interrupt their sitting.

During each activity regimen, participants will be asked to record all of the activities in an activity logbook. In addition, they will be asked to weigh (using kitchen scales) and record food and beverage consumption in a diary for the first four days (days 1-4) and then replicate the dietary intakes and timings exactly for the second four days (days 8-11). They will need to make sure that each meal contains at least 50% carbohydrate. Kitchen scales and a food diary will be provided by the research team.

Throughout the 11 days, participants will be required to avoid alcohol consumption and performing exercise (e.g. brisk walking, sports, going to the gym, cycling, running etc).

ELIGIBILITY:
Inclusion Criteria:

* Self-identified South Asian ethnicity.
* Self-report sitting at least 7 hours per day.
* Overweight or obese

Exclusion Criteria:

* Unable to speak and read English.
* Not able to performing light-intensity activities.
* Diagnosed cardiovascular disease or diabetes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 16 (Estimated)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Glycaemia | Net incremental area under the curve for interstitial glucose concentration during each 4-day condition will be calculated (i.e., the time frame is during the intervention)
  Net incremental area under the curve for each 4-day condition will be measured in the interstitial fluid of the subcutaneous tissue every minute and data averaged for each 15-min period will be stored and transmitted to a reader. The reader will be downloaded by the research team at the end of the last condition day.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bedfordshire, Bedford, Bedfordhsire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dey KC, Zakrzewski-Fruer JK, Smith LR, Jones RL, Maylor BD, Yates TE, Bailey DP. Substituting sitting with standing and walking in free-living conditions improves daily glucose concentrations in South Asian adults living with overweight/obesity. Eur J Appl Physiol. 2025 Aug 5. doi: 10.1007/s00421-025-05919-7. Online ahead of print. PMID 40764840